CLINICAL TRIAL: NCT00498199
Title: Visual Impairment, Oscillopsia and Multiple Sclerosis
Status: Terminated | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Other Study IDs: 2006.432
Record Dates: First submitted 2007-07-06; First posted 2007-07-09 (Estimated); Last update posted 2010-09-30 (Estimated); Status verified 2007-07

CONDITIONS: Multiple Sclerosis
Keywords: Multiples sclerosis; oscillopsia; eye movements; motion detection; retinal slip; nystagmus
MeSH Terms: conditions — Multiple Sclerosis; Nystagmus, Pathologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: visual tests

SUMMARY:
This study consists of two parts. The first part is a survey to examine vision-specific health-related quality of life in a cohort of patients with multiple sclerosis. We test visual impairment like visual acuity, visual field, colour discrimination, contrast sensitivity, eye movement. The aim of this part is to examine the association between responses to the quality of life scale and objective measures of visual impairment.

The second part is an open controlled study, in which we measure motion detection threshold in MS patients with oscillopsia due to pendular nystagmus and in a group of control subjects. The objective of this part is to determine whether patients with pendular nystagmus develop adaptation to oscillopsia using increased threshold of motion detection. We plan to test the effect of visuo-motor rehabilitation on this threshold in patients with oscillopsia due to pendular nystagmus.

DETAILED DESCRIPTION:
In the first part, 100 patients with multiple sclerosis are included. A vision-specific health-related quality of life scale and neuro-ophthalmological tests are administered. The duration of intervention is about 3 hours by patient and one year to finish this part.

In the second part, we include about 40 of 100 MS patients who present an oscillopsia due to pendular nystagmus and a group of 20 control subjects. The patients and subject will perform a motion detection task and the vision-specific health-related quality of life, the intervention lasting 1 hour. Then the patients will be randomized in one group treated by rehabilitation (one 30 mn session per week during 3 months) and the other one without treatment. A motion detection task and the vision-specific health-related quality of life scale will be performed at the end of the treatment for both groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 90
* Patients with established multiple sclerosis
* Visual impairment recovering from MS
* Understanding rules task
* Patient can stay set a long time
* Patient's agreement
* Membership to the Social Security
* No relapsing since three months

Exclusion Criteria:

* Brain damage
* Cognitive or behaviour disorder
* Patients with peripheral vestibular, otologic or ophthalmologic pathology antecedent
* Not stabilized disease (other one than MS)
* Patient under guardianship

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with established multiple sclerosis
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-04

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Tilikete, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Caroline Tilikete, Lyon, France